CLINICAL TRIAL: NCT02766452
Title: The Effects of a Preoperative Educational DVD on Parents' Participation in Their Child's Care in the Recovery Room at the Time of a Same-day Surgery: A Randomized Controlled Trial
Brief Title: Effects of Preparing Parents To Participate In Their Child's Care In The Recovery Room
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Collaborators: Children's Hospital of Eastern Ontario (Other)
Responsible Party: Principal Investigator, Julie Chartrand, Assistant Professor, University of Ottawa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 11/55X
Record Dates: First submitted 2016-05-05; First posted 2016-05-09 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: Perioperative Nursing

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pre-operative educational DVD preparation (Experimental): After their pre-assessment clinic (PAC) appointment, parents in the intervention group took the hospital's 20 minute surgical virtual tour in the hospital's family library. Parents in the intervention group also watched the 12 minute DVD entitled, "You and Your Child in the RR". This pre-operative educational tool was developed and tested in a previous study (Chartrand 2014). It was designed to enable parents to gain knowledge about the equipment and procedures related to the RR, and about nurses' and parents' roles in supporting their child in the RR. The DVD also focused on potential reactions of children waking up after a general anesthesia and strategies parents can use to support their child in the RR. The DVD included images of RR equipment and positive nurse-family and parent-child interactions.
  Interventions: Behavioral: "You and your child in the recovery room" DVD; Behavioral: Standard pre-operative preparation
- Standard pre-operative preparation (Placebo Comparator): After their PAC appointment, parents in the control groups took the hospital's 20 minute surgical virtual tour in the hospital's family library.
  Interventions: Behavioral: Standard pre-operative preparation

INTERVENTIONS:
Behavioral: "You and your child in the recovery room" DVD
  Arms: Pre-operative educational DVD preparation
Behavioral: Standard pre-operative preparation — Attendance to the Pre-anesthetic assessment clinic to meet with registered practical nurse and anesthesiologist (physical assessment and medical history). Completion of the Surgery Virtual Tour.

SUMMARY:
The objectives of this study were to evaluate the effect of a preoperative educational DVD on parents' knowledge acquisition, participation and anxiety related to their child's care in the recovery room (RR). It also aimed at evaluating the DVD in terms of children's postoperative distress, pain, analgesic requirements and length of recovery.

DETAILED DESCRIPTION:
Following the development of a validated preoperative educational Digital Versatile Disc (DVD) for parents, a randomized clinical trial, with a pre-test-post-test control group, was conducted on 123 French or English speaking parent-child dyads whose child was aged from 3 to 10 years and underwent an ear-nose-throat (ENT) or dental same day surgery at a Canadian pediatric hospital. The parents in the control group received the standard preoperative preparation (verbal and written information about hospital procedures and the hospital's surgical virtual tour). The parents in the experimental group viewed the DVD and received the standard preoperative preparation. Parents and children were videotaped in the recovery room; parental participation and children's distress were measured using observational scales. A validated multiple choice questionnaire was used to measure parents' knowledge acquisition, whereas a visual analogue scale allowed parents to report their anxiety level prior to, during and after their stay in the recovery room. A chart review was conducted to collect data on children's postoperative pain, analgesic requirements and length of recovery. In order to assess the effect of the DVD on parents and their child, T-test, chi-square analyses and repeated measures ANOVAs were conducted among 105 dyads.

ELIGIBILITY:
Inclusion Criteria:

* Parents speaking, reading and communicating to their child in english or french
* Parents who consented to participating in the study
* Parents who had a child aged 3 to 10 years who underwent a day surgery of the ENT type (an adenoidectomy or an amygdalectomy or a combination of both) or of the dental type (a dental exam under general anesthesia or an extraction or a dental repair under general anesthesia) were part of the sampling

Exclusion Criteria:

* The parents and the children who did not fit the eligibility criterias were excluded from the study.
* The parents who completed the consent form and questionnaires before the day of the surgery and who did the pre-surgical preparation, but who did not accompany the child in the recovery room were not part of the study.
* Also excluded, children who presented post-anesthetic complications (ex.: respiratory distress, hemorrhage, severe emotional distress, etc.).
* Children presenting surgical complications (ex.: cardio-respiratory distress and hemorrhage) were also excluded from the study.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2011-09; Primary Completion 2012-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Parents' participation behaviors | Post-treatment (In average, between 1 and 7 days following the intervention)
  Video recordings were taken of parents and children during the child's stay in the recovery room, every 3 minutes for 15 seconds at a time. A maximum of six segments were randomly selected to capture a range of parental participation behaviors throughout their stay in the RR. Thus, the maximum duration of the recordings was 1 ½ minutes per parent (six observation periods x 15 seconds). Parents' participation behaviors were measured using an observational checklist, the Inventaire des conduites parentales (ICP) (Parental Behaviours Inventory), which includes different behaviors parents may have during a child's same-day surgery (Tourigny et al., 2005). The ICP is composed of 13 indicators divided into three categories; verbal information (i.e. providing information to child and answering child's questions), cognitive strategies (i.e. applying positive reinforcement and implementing coping strategies) and attitudes (i.e. showing the child affection and being close to the child).

SECONDARY OUTCOMES:
Parents' knowledge acquisition | Post-treatment (In average, between 1 and 7 days following the intervention)
  A multiple choice questionnaire was designed and validated for this study, then used to measure parents' knowledge. Parents' answers were tabulated to get a total score for each parent and for each test (test 1: Pre-intervention and test 2: Post-intervention). The maximum score for each test was 10. Parents' knowledge acquisition was measured by calculating the difference between parents' scores on test 1 and test 2.
Parents' anxiety | Post-treatment (In average, between 1 and 7 days following the intervention)
  Defined by parents' self-reporting of their anxiety at three time points: 1) immediately before entering the RR; 2) 5 minutes after entering the RR; and 3) 5 minutes after leaving the RR with their child. Parents' anxiety was measured using the Visual Analogue Scale for Anxiety (VAS-A) (Vogelsang 1988)
Children's distress in the recovery room (RR) | Post-treatment (In average, between 1 and 7 days following the intervention)
  Defined as facial, verbal, and affective manifestations, and motor indicators of emotional distress related to anxiety, anger, fear and pain. Parent-child dyads were digitally video-recorded in the RR. The video segments randomly selected to measure parents' participation behaviours in the RR were also used to measure children's distress behaviours. Children's distress behaviours were measured with the Échelle descriptive du comportement de l'enfant opéré (EDCEO) (Observation scale to assess the behaviour of children undergoing surgery) (Tourigny 2000)
Children's pain | Post-treatment (In average, between 1 and 7 days following the intervention)
  Post-operative pain was assessed in the RR and the daycare surgery (DCS) unit and documented by nurses using the Modified Children's Hospital of Eastern Ontario Pain Score (mCHEOPS) (Splinter et al. 1994)
Children's analgesic requirements | Post-treatment (In average, between 1 and 7 days following the intervention)
  Post-operative analgesics required by children in the RR and in the DCS unit included opioid analgesics (e.g. Fentanyl and Morphine) and non-opioids (e.g.
  Acetaminophen)
Children's length of recovery | Post-treatment (In average, between 1 and 7 days following the intervention)
  Time (in minutes) elapsed between the arrival of the children in the RR and their departure from the DCS unit. The time at which children were discharged from the DCS unit was determined based on the achievement of specific criteria regarding level of activity and consciousness, vital signs, blood perfusion, pain and wound assessment and feeding.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tourigny J, Chapados C, Pineault R. Determinants of parental behaviour when children undergo day-care surgery. J Adv Nurs. 2005 Dec;52(5):490-7. doi: 10.1111/j.1365-2648.2005.03617.x. PMID 16268854
- [Background] Vogelsang J. The Visual Analog Scale: an accurate and sensitive method for self-reporting preoperative anxiety. J Post Anesth Nurs. 1988 Aug;3(4):235-9. No abstract available. PMID 2457102
- [Background] Tourigny J. [A new instrument to measure distress in the operated child]. Infirm Que. 2000 Nov-Dec;8(2):18-26, 28-9. French. PMID 11885458
- [Background] Splinter, W. M., Semelhago, L. C., et Chou, S. (1994). The reliability and validity of a modified CHEOPS pain score. Anesthesia and Analgesia, 78, S413.
- [Result] Chartrand, J. (2014). Effet d'un DVD éducatif pré-opératoire sur les connaissances et les conduites des parents en salle de réveil: une étude clinique randomisée (Doctoral dissertation, Université d'Ottawa). Retrieved from http://hdl.handle.net/10393/31231
- [Derived] Chartrand J, Tourigny J, MacCormick J. The effect of an educational pre-operative DVD on parents' and children's outcomes after a same-day surgery: a randomized controlled trial. J Adv Nurs. 2017 Mar;73(3):599-611. doi: 10.1111/jan.13161. Epub 2016 Oct 20. PMID 27681601